CLINICAL TRIAL: NCT04153214
Title: Effects of Cycling Workstation on Cardiometabolic Health for Workers With an Office-sitting Desk
Brief Title: Effects of Cycling Workstation on Cardiometabolic Health for Workers With an Office-sitting Desk (REMOVE)
Acronym: REMOVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire AME2P - Unversité Clermont Auvergne (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2019 DUCLOS 2; 2019-A04449-48 (Other: ANSM)
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Sedentary Behavior
Keywords: Cardiometabolic health; Sedentary Behavior; Active workstation; Cycling desk
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycling workstation (Experimental): Participants will have a portable pedal machine under their desk and will use it 60minutes per day (30minutes in the morning and 30minutes in the afternoon) during 6 months
  Interventions: Behavioral: cycling
- control (Placebo Comparator): Daily activities unchanged during 3 months. Then they will have a portable pedal machine under their desk and will use it 60minutes per day (30minutes in the morning and 30minutes in the afternoon) during 3 months.
  Interventions: Behavioral: cycling

INTERVENTIONS:
Behavioral: cycling — Participants will have a portable pedal machine under their desk and will use it 60minutes per day

SUMMARY:
The recent literature has highlighting the importance of the time of inactivity and the level of physical activity (PA) as predictors of metabolic cardio risks. Now, sedentary lifestyles are well recognized as one of the causes of mortality. As with physical activity, a dose-response relationship appears to exist: mortality would increase with time spent in sedentary behaviors. However, this relationship would not be linear: the more the daily sitting time increases, the more the consequences on mortality are important. It is now well demonstrated that time spent in sedentary adult behaviour finds primarily its origin in the work, characterized by prolonged and uninterrupted periods of sitting. Many strategies have been settled to break the prolonged sitting time. The most promising one seem to be the use of active workstations (treadmill, cycling, stepping) because they reduce sedentary time at work and increase physical activity with positive effects on the global health. If active workstations have demonstrated their effectiveness with overweight or obese people by increasing daily energy expenditure, their interest in prevention in normal weight people is less known. In addition, the long-term effectiveness of a program of reactivation by active workstation on biological parameters, quantitative and qualitative time of sedentary behaviour (duration, number of breaks) and physical fitness was not assessed.

The main objective of this project is to study the effects of the use of a cycling workstation for 60 minutes per day (30 minutes twice a day) for 3 months among professionals with an office-sitting desk on overall quantity of physical activity time (work and non-work) and sedentary time.

DETAILED DESCRIPTION:
Subject will have a pre-inclusion visit during a medical consultation where the eligibility criteria to participate to this study will be checked.

After the inclusion of subject and their agreements to participate to the study, they will know in which group they are :

* Group who performs 30minutes twice a working day from day 1 to day 180 (interventional)
* Group who performs 30minutes twice a working day from day 90 to day 180 (control)

They will have evaluation at three different times : T0 (Day 1), T1 (Day 90), T2 (Day 180). The evaluation will evaluate :

* overall quantity and quality of physical activity time (work and non-work) and sedentary time
* Body composition
* Biological parameters
* Physical fitness
* Psychological parameters At the end of the protocol, there will be an assessment of the obstacles or motivations to this program.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer, male or female, between 18 and 61 years old
* Body mass index > 18,5 kg/m2 and ≤ 35 kg/m2
* More than 0.8 full time equivalent hours (FTE) with 75% of this time in a sitting position
* Able to provide informed consent to research participation
* Registered in the French social security system

Exclusion Criteria:

* Work involving multiple periods of sitting interruptions >1 minute
* Subject using a sit-to-stand office desk or a swiss ball
* Sports activity > 2.5 hours/week
* Contact jobs (face-to-face with people)
* Pregnant or breastfeeding women
* Medical or surgical history determined by principal investigator to be not compatible with the study
* Subject with cardiorespiratory and/or osteo-articular disorders limiting their ability to perform physical tests or the use of active offices
* Subject with type 1 or type 2 diabetes treated with insulin
* Subject with progressive cardiovascular or neoplastic disease.
* Subject with a major infection within 3 months of inclusion.
* Subject with known neuromuscular pathology: myopathy, myasthenia, rhabdomyolysis, paraplegia, hemiplegia
* Subject with chronic or acute inflammatory pathology 3 months prior to inclusion
* Subject treated by beta-blocker
* Subject diagnosed and/or treated for schizophrenia, bipolar disorders, major depression
* Subject treated, or having stopped treatment for less than 3 months prior to inclusion, by corticosteroids, immunosuppressant, anabolic, growth hormone.
* Subject with unstable psychiatric condition
* Significant alcohol consumption (> 2-3 drinks per day depending on gender) or presence of substance abuse.
* Unable to walk or pedal 45 minutes in a row
* Subject who is excluded from another study or who received more than €4,500 in the year following his participation in clinical studies
* Subject deprived of their liberty by judicial or administrative decision
* Refusal to sign written consent to participate
* Subject participating in another study

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
effects of the use of a cycling Workstation for 60 minutes per day (30 minutes twice a day) for 3 months among professionals with an office-sitting desk on overall quantity of physical activity time (work and non-work) and sedentary time | month 3
  Quantify by the use of an accelerometer device wears at the hip

SECONDARY OUTCOMES:
Body composition | day 90
  Body fat mass, body fat free mass will be assessed by bioimpedance analysis
Body composition | day 180
  Body fat mass, body fat free mass will be assessed by bioimpedance analysis
Body composition | day 1
  Body fat mass, body fat free mass will be assessed by bioimpedance analysis
Biological parameters - insulin | Day 1
  will be assessed in the fasting state using blood sample (insulin mlUI/L)
Biological parameters - insulin | Day 90
  will be assessed in the fasting state using blood sample (insulin mlUI/L)
Biological parameters - insulin | Day 180
  will be assessed in the fasting state using blood sample (insulin mlUI/L)
Biological parameters - glucose | Day 1
  will be assessed in the fasting state using blood sample (glucose g/L)
Biological parameters - glucose | Day 90
  will be assessed in the fasting state using blood sample (glucose g/L)
Biological parameters - glucose | Day 180
  will be assessed in the fasting state using blood sample (glucose g/L)
Biological parameters - triglycerides | Day 1
  will be assessed in the fasting state using blood sample (triglycerides g/L)
Biological parameters - triglycerides | Day 90
  will be assessed in the fasting state using blood sample (triglycerides g/L)
Biological parameters - triglycerides | Day 180
  will be assessed in the fasting state using blood sample (triglycerides g/L)
Biological parameters - cholesterol | Day 1
  will be assessed in the fasting state using blood sample (cholesterol g/L)
Biological parameters - cholesterol | Day 90
  will be assessed in the fasting state using blood sample (cholesterol g/L)
Biological parameters - cholesterol | Day 180
  will be assessed in the fasting state using blood sample (cholesterol g/L)
Biological parameters - CRP | Day 1
  will be assessed in the fasting state using blood sample (CRP-us mg/L)
Biological parameters - CRP | Day 90
  will be assessed in the fasting state using blood sample (CRP-us mg/L)
Biological parameters - CRP | Day 180
  will be assessed in the fasting state using blood sample (CRP-us mg/L)
Biological parameters - anandamide | Day 1
  will be assessed in the fasting state using blood sample (plasma concentration anandamide pmol/ml)
Biological parameters - anandamide | Day 90
  will be assessed in the fasting state using blood sample (plasma concentration anandamide pmol/ml)
Biological parameters - anandamide | Day 180
  will be assessed in the fasting state using blood sample (plasma concentration anandamide pmol/ml)
Psychological assessment | Day 1
  Through an evaluation of healthy life span, stress at work and outside, stress management and anxiety (questionnaires)
Psychological assessment | Day 90
  Through an evaluation of healthy life span, stress at work and outside, stress management and anxiety (questionnaires)
Psychological assessment | Day 180
  Through an evaluation of healthy life span, stress at work and outside, stress management and anxiety (questionnaires)
Resting metabolic rate | Day 1
  will be assessed at rest during 30 minutes using indirect calorimetry
Resting metabolic rate | Day 90
  will be assessed at rest during 30 minutes using indirect calorimetry
Resting metabolic rate | Day 180
  will be assessed at rest during 30 minutes using indirect calorimetry
Physical capacity | Day 1
  will be assessed with the Step Test 6 minutes
Physical capacity | Day 90
  will be assessed with the Step Test 6 minutes
Physical capacity | Day 180
  will be assessed with the Step Test 6 minutes
Muscle Strength | Day 1
  will be assessed with handgrip for upper limb muscle and isokinetic dynamometer for lower limb muscle
Muscle Strength | Day 90
  will be assessed with handgrip for upper limb muscle and isokinetic dynamometer for lower limb muscle
Muscle Strength | Day 180
  will be assessed with handgrip for upper limb muscle and isokinetic dynamometer for lower limb muscle
Quality of the time spend to physical activities and sedentary behaviour | Day 1
  * moderate and high intensity physical activity
  * low intensity physical activity
  * total sedentary time
  * number of sedentary periods of ≥30 minutes, ≤10 minutes, 10 to 30 minutes Evaluate by the use of an accelerometer device wears at the hip
Quality of the time spend to physical activities and sedentary behaviour | Day 90
  * moderate and high intensity physical activity
  * low intensity physical activity
  * total sedentary time
  * number of sedentary periods of ≥30 minutes, ≤10 minutes, 10 to 30 minutes Evaluate by the use of an accelerometer device wears at the hip
Quality of the time spend to physical activities and sedentary behaviour | Day 180
  * moderate and high intensity physical activity
  * low intensity physical activity
  * total sedentary time
  * number of sedentary periods of ≥30 minutes, ≤10 minutes, 10 to 30 minutes Evaluate by the use of an accelerometer device wears at the hip

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Nasir H, Dutheil F, Ramos I, Guirado T, de Saint-Vincent S, Thivel D, Metz L, Duclos M. Effects of portable pedal machines at work on lipoprotein subfraction profile in sedentary workers - the REMOVE study. Lipids Health Dis. 2024 Apr 14;23(1):105. doi: 10.1186/s12944-024-02098-w. PMID 38616275
- [Derived] Guirado T, Metz L, Pereira B, Brun C, Birat A, Boscaro A, Bergouignan A, Thivel D, Duclos M. A 12-Week Cycling Workstation Intervention Improves Cardiometabolic Risk Factors in Healthy Inactive Office Workers. J Occup Environ Med. 2022 Aug 1;64(8):e467-e474. doi: 10.1097/JOM.0000000000002583. Epub 2022 Jun 11. PMID 35673701
- [Derived] Guirado T, Metz L, Pereira B, Bergouignan A, Thivel D, Duclos M. Effects of cycling workstation to get tertiary employee moving on their overall health: study protocol for a REMOVE trial. Trials. 2021 May 22;22(1):359. doi: 10.1186/s13063-021-05317-2. PMID 34022938